CLINICAL TRIAL: NCT03516838
Title: Clinical and Radiographic Evaluation of a New Bioactive Ionic Resin Material (ACTIVA™ BioACTIVE) Versus Compomer for Class II Restorations in Primary Molars: A Split Mouth Randomized Clinical Trial
Brief Title: Comparison of ACTIVA BioACTIVE Versus Compomer in Restoring Dental Decay in Primary Molar Teeth
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EC UZG 2016/1050 - 1051
Record Dates: First submitted 2018-04-22; First posted 2018-05-04 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Dental Caries in Children
Keywords: Dental caries; Class II; Primary molar; Restorative material; Bioactive material; Compomer; Activa bioactive; Ryge criteria
MeSH Terms: conditions — Dental Caries | interventions — Compomers; Dyract

STUDY DESIGN:
Intervention Model Description: Experimental prospective double blinded split-mouth randomized controlled trial .
  Each patient receive both types of treatment in the oral cavity, one type of the treatment on each side.
  The patients act as their control
Who Masked: Participant, Outcomes Assessor
Masking Description: During treatment, the type of filling material was concealed from the patient, and the patient had no information which material was used in each side of the mouth. The type of material was not mentioned in the patient's file. Instead, it was replaced by a combination which the outcomes assessors were not familiar with. The operator was also blinded for the type of restoration during tooth preparation and was informed only at the time of restoration placement. The purpose of this discretion was to ensure double blinding both at the patient, as well as the outcomes assessor level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ACTIVA™ BioACTIVE (Experimental): Restoring cavity using ACTIVA filling material
  Interventions: Drug: ACTIVA™ BioACTIVE
- Compomer (Active Comparator): Restoring cavity using compomer filling material
  Interventions: Drug: Compomer

INTERVENTIONS:
Drug: ACTIVA™ BioACTIVE — Restorative Dental Material: Permanent resin containing filling dental material with bioactive properties to restore decayed teeth
  Other Names: ACTIVA
  Arms: ACTIVA™ BioACTIVE
Drug: Compomer — Restorative Dental Material: Permanent resin containing filling dental material to restore decayed teeth
  Other Names: Dyract
  Arms: Compomer

SUMMARY:
A clinical trial to evaluate a filling material (ACTIVA) and compare it to a traditional filling material (compomer) to restore decayed deciduous teeth in children

DETAILED DESCRIPTION:
A tooth decay in deciduous teeth has to be restored with proper filling material. ACTIVA™ BioACTIVE is a new filling material which has the ability to release and recharge fluoride in the oral cavity which is important for preventing further tooth decay. In this study we will compare this new filling material with Compomer (the traditional control filling material) by restoring decayed deciduous molars with one of the mentioned filling materials.

Both filling materials have no reported adverse effect and used regularly in the dental practice.

The treatment procedure is performed in healthy children from both genders with decayed deciduous molars aged between 5 to 10 years by one operator in the dental chair under local anesthesia in the department of pediatric dentistry and special care, Ghent University hospital, Ghent, Belgium.

At least 35 teeth is needed to demonstrate an effect. Each material is placed randomly based on randomization done by the computer. Each participant will receive both types of treatments, one type on each side of the mouth.

The participants will come back each six months to check the success of each treatment group by two trained dentists other than the operator. and to check whether the control group performs similar, better or worse than the control group.

The duration of treatment procedure of both treatment groups is recorded and compared to check if one filling material takes less time than the other to placed in the oral cavity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children with American Society of Anesthesiologists (ASA) I score from both gender aged between three and ten years
* Vital decayed deciduous molar with proximal enamel/dentine caries
* At least one decayed tooth on each side of the mouth (split mouth)
* Pt is treatable in the dental chair
* Parents agreed to participate in the study and signed the informed consent

Exclusion Criteria:

* Patients with medical conditions or systemic disease
* Anxious or uncooperative patients who are not treatable in the dental chair
* Any symptoms like: pain, swelling, abscess or fistula.
* Extensive caries, dental developmental disturbance, pathological mobility, pulp exposure or indication for pulp therapy
* Patients with one decayed tooth in the whole mouth (not split mouth)

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation | 6 months follow-up
  Check the filling clinically based on United States Public Health Ryge criteria by a blinded and calibrated assessor
Clinical evaluation | 12 months follow-up
  Check the filling clinically based on United States Public Health Ryge criteria by a blinded and calibrated assessor
Radiographic evaluation | 12 months follow-up
  Check the filling radiographically based on Rx photo by a blinded and calibrated assessor

SECONDARY OUTCOMES:
Time needed to place the filling material | Immediately after each intervention
  Time since start placing the filling material until finishing the restoration is recorded and compared between the two groups to investigate whether both materials take the same time to be placed in the oral cavity.

CONTACTS AND LOCATIONS:
Overall Officials: Luc Martens, PhD, Study Director — PaeCoMeDis Research group,Ghent University Hospital
Locations (1):
- Ghent University hospital, Ghent, Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data will be available in the literature in the manuscript after publication
Supporting Information: Study Protocol, SAP
Time Frame: After publication

REFERENCES:
- [Derived] Banon R, Vandenbulcke J, Van Acker J, Martens L, De Coster P, Rajasekharan S. Two-year clinical and radiographic evaluation of ACTIVA BioACTIVE versus Compomer (Dyract(R) eXtra) in the restoration of class-2 cavities of primary molars: a non-inferior split-mouth randomised clinical trial. BMC Oral Health. 2024 Apr 10;24(1):437. doi: 10.1186/s12903-024-04132-w. PMID 38600533